CLINICAL TRIAL: NCT00374049
Title: A Pilot Dose Finding Study of MUC1 Vaccine in Conjunction With Poly-ICLC (Polyinosinic-polycytidylic Acid Stabilized With Polylysine and Carboxymethylcellulose) or HiltonolTM in Patients With Recurrent and/or Advanced Prostate Cancer
Brief Title: MUC1 Vaccine in Conjunction With Poly-ICLC in Patients With Recurrent and/or Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Olivera Finn (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Olivera Finn, Distinguished Professor and Chair, Department of Immunology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-086
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
Keywords: Prostate; vaccine; immunosuppression; dendritic cells
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One (Experimental): MUC1 vaccine in conjunction with GM-CSF and Poly-ICLC (Hiltonol)in Arm ONE
  Interventions: Drug: MUC_1

INTERVENTIONS:
Drug: MUC_1 — Pretreatment with Poly-ICLC alone week 1 &2 (50 ug/kg 3 days/week) Weeks 3-7 Poly-ICLC, 2 days/week; MUC-1 vaccine (100ug) admixed with GM-CSF (100ug), administered subcutaneously at weeks 3, 5 and 7 Tetanus toxoid, administered via intramuscular injection, 1x at week 3 GM-CSF 100ug, administered subcutaneously on days 2-4

SUMMARY:
The purpose of this study is to determine the effectiveness of a drug called Poly-ICLC, also known as HiltonolTM, in boosting the body's immune system's response to an experimental vaccine therapy (called the MUC-1 vaccine).

DETAILED DESCRIPTION:
This is a one-arm clinical trial, to evaluate 2 doses of poly-ICLC for reversing systemic immuno-suppression: 25 μg/kg and 50 μg/kg. These doses will be administered I.M. three times a week for 2 weeks. Following 2 weeks of treatment with poly-ICLC alone, patients will be immunized subcutaneously with the 100-mer MUC-1 peptide + GM-CSF. Subjects will be boosted twice at two week intervals, and subsequently 3 months later, if they experience clinical benefit or if they have clinically stable disease. Poly-ICLC will be administered continually 3 times a week I.M. for the first 2 weeks and 2 times a week I.M. thereafter. Subjects will continue on study until they have evidence of progressive disease. The primary objective of this study is to evaluate the efficacy of Poly-ICLC in boosting the immunologic response of a MUC1 vaccine. Secondary objectives are to evaluate a) changes in markers of systemic immunosuppression; b) changes in dendritic cell number and function; and c) clinical response. Up to 30 subjects will be enrolled in this single-site study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and must have histologically confirmed adenocarcinoma of the prostate with systemic disease are potentially eligible. Patients with an early relapse must have undergone and failed definitive surgery and/or radiation. Patients can either be hormone naive, may be on concurrent hormone therapy with LHRH analogues, or may be hormone refractory (see section 3.1.4 of the full protocol)
* Must have evidence of systemic immunosuppression as evidenced by the presence of one or more of the following: 1) Low or absent T cell zeta chain expression in peripheral blood (PB), 2) Low level cytokine production ( i.e., IFN-gamma , IL-4 ) by T cells in PB, 3) Upregulation of granulocyte activation markers (CD 15) in PB
* Availability of at least 2 PSA measurements over 2 to 6 weeks, clearly documenting a rising PSA. The minimum rise in PSA must be at least 50% from baseline PSA. The last of these PSA values must be > 2 .
* Patients may be hormone-refractory (rising PSA, despite castrate testosterone levels, i.e., < 50 ng/ml); may have metastatic disease; and maybe on bisphosphonates. If patients are on anti-androgens (Flutamide/Casodex), they must have been off of these agents for at least 28 days prior to enrollment for flutamide, and at least 42 days prior to enrollment for bicalutamide (Casodex)), without a drop in PSA. If hormone refractory, patients will continue LHRH analogues.
* Signed written informed consent given by the patient before or at enrollment in the study and following receipt of verbal and written information about the study.
* No concomitant therapy with steroids
* No other investigational therapy within 4 weeks of enrolling on this protocol
* No chemotherapy or radiation therapy within 6 weeks of enrolling on this protocol.
* ECOG performance status 0 or 1
* Patients must have adequate organ and marrow function
* Men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients who have had chemotherapy or radiation therapy within 6 weeks of study entry.
* No concurrent use of other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Presence of an active acute or chronic infection, including urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology). HIV patients are excluded based on immunosuppression which may render them unable to respond to the vaccine; patients with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Patients with either previously irradiated or new CNS (central nervous system) metastases at entry are excluded. Pre-enrollment head CT is not required if not indicated by clinical signs or symptoms.
* Patients with a history of auto-immune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* Subjects with active prior malignancy within the past 5 years (with exception of non-melanoma skin cancers and carcinoma in situ of the bladder).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing an immunologic response at week 8 | 8weeks

SECONDARY OUTCOMES:
Measures of systemic immunosuppression | 8weeks
Dendritic cell (DC) status | 7 weeks
T cell subset analyses | 8weeks
Clinical Response | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States